CLINICAL TRIAL: NCT05656248
Title: A Prospective,Single Site, Single-Arm Pilot Study of CPX-351 (VYXEOS) in Individuals < 22 Years With Secondary Myeloid Neoplasms
Brief Title: Study of CPX-351 (VYXEOS) in Individuals < 22 Years With Secondary Myeloid Neoplasms
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPXSMN; NCI-2022-10271 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-10

CONDITIONS: Myeloid Neoplasm
Keywords: Acute myeloid leukemia (AML); Myelodysplastic syndrome (MDS); Chronic myelomonocytic leukemia (CMML)]
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Juvenile | interventions — CPX-351; Cytarabine; Daunorubicin; Methotrexate; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CPX-351 (Experimental): Participants will receive CPX-351 for remission induction, and then will proceed to allogeneic HSCT or other therapies as per institutional practice.
  Intrathecal (IT) chemotherapy will be given on Day 1 of each cycle, for all participants, but may be delayed if clinically indicated. IT cytarabine, IT methotrexate, and IT methotrexate/hydrocortisone/cytarabine (MHA) according to age are all acceptable.
  Interventions: Drug: CPX-351; Drug: MHA; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation

INTERVENTIONS:
Drug: CPX-351 — Given Intraveneously (IV)
  Other Names: Vyxeos®; cytarabine/daunorubicin liposomal
Drug: MHA — Given Intrathecal (IT)
  Other Names: methotrexate/hydrocortisone/cytarabine
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo HSCT
  Other Names: HSCT; Stem Cell Transplantation

SUMMARY:
The purpose of this study is to learn the effects of treatment with an investigational drug, CPX-351 in patients with secondary myeloid neoplasms (SMNs).

DETAILED DESCRIPTION:
Primary Objective

* Determine the composite complete remission (CR) and complete remission with incomplete peripheral blood recovery (CRi) rates, safety and tolerability in patients under 22 years of age with SMN treated with one or two courses of CPX-351 before HSCT.

Secondary Objectives

* Describe the toxicity profile of patients with SMN treated with one or two courses of CPX-351.
* Describe the biologic correlates of response in patients with SMN after one or two courses of CPX-351.
* Estimate the 3-year overall survival of patients who received one or two courses of CPX-351 followed by HSCT.

Participants who meet the inclusion criteria and consent will receive up to 2 cycles of CPX-351 for remission induction, and then will proceed to allogeneic HSCT or other therapies as per institutional practice. If a patient attains remission and has negative MRD after the first course of CPX-351, and HSCT can occur within 3 to 4 weeks from the evaluation date of the first course, the patient can proceed to HSCT without receiving the second course of CPX-351.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥1 year and < 22 years of age at the time of enrollment.
* Patient must have one of the following diagnoses:

  * Treatment-related MDS/AML: Patients with solid organ or hematopoietic neoplasms previously treated with alkylating agents, ionizing radiation, topoisomerase inhibitors, antimetabolites, thiopurines, mycophenolate mofetil, fludarabine, and anti-tubulin agents (vincristine, vinblastine, vindesine, paclitaxel, and docetaxel usually in combination), who develop MDS, or AML are candidates for the CPXSMN protocol. If the bone marrow has between 5% and 20% blasts (higher-risk MDS), patients are discussed with the hematopoietic stem cell transplantation (HSCT) team for consideration to receive chemotherapy before HSCT. If the consensus is that cytoreduction before HSCT is necessary, and the cumulative dose of doxorubicin equivalent is < 500 mg/m2 (in cases of cardio protection) or ≤400 mg/m^2 (cases without cardio protection), patients are eligible for the CPXSMN protocol OR
  * Secondary MDS/AML: Patients with primary MDS in transformation to AML (refractory cytopenia with an excess of blasts), acquired aplastic anemia evolving to AML, myeloid neoplasms arising from inherited bone marrow failure syndromes (including severe congenital neutropenia, Schwachman-Diamond syndrome, MECOM syndrome) or MDS/AML predisposition syndromes (including germline predisposition in GATA2, RUNX1, SAMD9/SAMD9L, ERCC6L2, NF1, ETV6, ANKRD26, ERCC6L2, TP53 or CEBPA genes) are eligible for the CPXSMN trial. If the bone marrow has between 5% and 20% blasts (higher-risk MDS), patients are discussed with the HSCT team for consideration to receive chemotherapy before HSCT. If the consensus is that cytoreduction before HSCT is necessary, the patients are eligible for the CPXSMN protocol.
* Patients must have a performance status corresponding to an Eastern Cooperative Oncology Group (ECOG) score of 0, 1 or 2. Use Karnowski for patients > 16 years of age and Lansky for patients ≤16 years of age.

  * Note: Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Concomitant medications restrictions

  * See Section 4.2.5 or Appendix II (of protocol) for concomitant therapy restrictions for patients during treatment.
* Adequate renal function defined as:

  * Creatinine clearance or radioisotope GFR > 70 mL/min/1.73 m^2, or
  * A serum creatinine based on age/gender as follows: Age: 1 to < 2 years; Maximum Serum Creatinine: Male 0.6, Female 0.6; Age: 2 to < 6 years, Maximum Serum Creatinine: Male 0.8, Female 0.8; Age: 6 to < 10 years; Maximum Serum Creatinine: Male 1, Female 1; Age: 10 to < 13 years; Maximum Serum Creatinine: Male 1.2, Female 1.2; Age: 13 to < 16 years; Maximum Serum Creatinine: Male 1.5, Female 1.5; Age: ≥ 16 years; Maximum Serum Creatinine: Male 1.7, Female 1.4
* Adequate liver function defined as (unless it is related to leukemic involvement):

  * Direct bilirubin ≤1.5 x upper limit of normal (ULN) for age and institution. At institutions that do not obtain a direct bilirubin in patients with a normal total bilirubin, a normal total bilirubin may be used as evidence that the direct bilirubin is not > 1.5 x the ULN.
  * SGPT (ALT) ≤ 3.0 x ULN for age and institution
* Adequate cardiac function defined as:

  * Shortening fraction of ≥27% by echocardiogram, or
  * Ejection fraction of ≥ 50% by radionuclide angiogram or echocardiogram, and
  * Corrected QT (QTcB) interval < 500 msecs
* Central nervous system function defined as:

  * Patients with seizure disorder may be enrolled if on anticonvulsants and if seizures are well controlled
  * CNS toxicity ≤ Grade 2
* Prior therapy

  * Patients must have recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, HSCT or radiotherapy prior to entering this study. All prior treatment-related toxicities must have resolved to ≤ Grade 2 prior to enrollment.

    1. Myelosuppressive chemotherapy: Must not have received myelosuppressive chemotherapy within 3 weeks of entry onto this study (excluding hydroxyurea). Cyto-reduction with hydroxyurea can be initiated and continued for up to 24 hours prior to the start of CPX-351.
    2. Biologic (anti-neoplastic agent): At least 7 days since the completion of therapy with steroids, retinoids or hypomethylating agents. Note: For agents that have known adverse events occurring beyond 7 days after administration (i.e. monoclonal antibodies), this period must be extended beyond the time during which acute adverse events are known to occur.
    3. Radiation therapy (RT): ≥ 2 weeks for local palliative RT (small port); ≥ 6 months must have elapsed if prior craniospinal RT or if ≥ 50% radiation of pelvis; ≥ 6 weeks must have elapsed if other substantial BM radiation. Note: Patients must have received ≤ than 13.6 Gy prior radiation to the mediastinum. Patients with prior cumulative doxorubicin equivalent > 400 mg/m2 and prior radiation (any dose) to the mediastinum are not eligible for the protocol.
    4. Hematopoietic stem cell transplantation: No evidence of active graft vs. host disease for at least 4 weeks. For allogeneic HSCT patients, ≥ 3 months must have elapsed since HSCT.

       * Must have received no more than 1 prior autologous or allogeneic stem cell transplant.
       * Patients must be off all systemic immunosuppressive therapy for at least 2 weeks, excluding hydrocortisone for physiologic cortisol replacement.
    5. Intrathecal cytotoxic therapy:

       * No waiting period is required for patients having received intrathecal cytarabine, methotrexate, and/or hydrocortisone.
       * At least 14 days must have elapsed since receiving liposomal cytarabine (DepoCyte) by intrathecal injection.
    6. Growth factors:

       * Patients must not have received hematopoietic growth factors for 7 days prior to CPX-351.
       * Patients must not have received pegfilgrastim for 14 days prior to CPX-351.
* HIV disease

  * Patients with a known history of HIV are eligible, if they meet all of the following conditions:

    * No history of HIV complications with the exception of CD4 count < 200 cells/mm^3
    * No antiretroviral therapy with overlapping toxicity such as myelosuppression
    * CD4 count > 500 cells/mm^3 prior to the diagnosis of relapsed AML
    * HIV viral loads below the limit of detection
    * No history of highly active antiretroviral therapy (HAART)-resistant HIV
* Residual or relapsed solid malignancy

Patients with residual or relapsed solid malignancy (for example osteosarcoma) at the time of the diagnosis of SMN are not excluded from this trial and the treatment individualized to integrate the management of the two malignancies.

* All patients and/or their parents or legal guardians must sign a written informed consent.

Exclusion Criteria:

* Patients with de novo AML (i.e., patients eligible for St. Jude or COG frontline AML trials).
* Patients with any of the following:

  * Constitutional trisomy 21 or with constitutional mosaicism of chromosome trisomy 21
  * Patients with Fanconi anemia (DNA repair syndrome) or dyskeratosis congenita (telomeropathy)
  * Wilson disease or other copper-related metabolic disorders
  * Mixed phenotype acute leukemia
  * Philadelphia chromosome-positive myeloid neoplasms (AML or CML)
  * Acute promyelocytic leukemia (APL), or
  * Juvenile myelomonocytic leukemia (JMML) and related RASopathy disorders in chronic phase.
* Patients who have received greater amount of doxorubicin equivalents to <500 mg/m2 (in cases of cardio protection with dexrazoxane) or <400mg/m2 (cases without cardio protection). For the purposes of determining eligibility for this protocol, the following cardiotoxicity multipliers will be used to determine doxorubicin equivalents:

  * Doxorubicin (reference): 1
  * Daunomycin: 0.5
  * Epirubicin: 0.5
  * Idarubicin: 5
  * Mitoxantrone: 10
* Patients who are currently receiving another investigational drug.
* Patients receiving medications for treatment of left ventricular systolic dysfunction.
* Patients with documented active, uncontrolled infection at the time of study entry.
* Patients with known active HBV and HCV infections.
* Patients with prior allergy to daunorubicin and/or cytarabine.
* Pregnancy and breast feeding

  * Female patients who are pregnant are ineligible due to risks of fetal and teratogenic adverse events as seen in animal/human studies.
  * Lactating females who are breastfeeding an infant/child
  * Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained.
  * Sexually active patients of reproductive potential are not eligible unless they have agreed to use an effective contraceptive method for the duration of their study participation and for at least 6 months after the last dose of protocol therapy.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Composite complete remission (CR) rates after one or two courses of CPX-351 | After one or 2 course of CPX-351, no later than day 42 from the start of each course of chemotherapy
  The Simon's two-stage minimax design with be used. Complete morphologic remission response (CR) is defined as less than 5% blasts without Auer rods by morphological evaluation of the bone marrow (M1 marrow).
Complete remission with incomplete peripheral blood recovery (CRi) rates after one or two courses of CPX-351 | After one or 2 course of CPX-351, no later than day 42 from the start of each course of chemotherapy
  The Simon's two-stage minimax design with be used. Complete remission with incomplete peripheral blood recovery (CRi) is defined as hematologic recovery hematological (white cell blood count ≥ 1.0 x 109/L, unsupported platelet count ≥ 30.0 x 109/L and absolute neutrophil count ≥ 0.3 x 109/L).
Safety and tolerability in patients under 22 years of age with SMN treated with one or two courses of CPX-351 before HSCT | After one or 2 course of CPX-351, prior to hematopoietic stem cell transplantation (HSCT), three to four weeks from the hematologic recovery
  The exact three-stage binomial design will be used to monitor tolerability. We define a tolerability success as a patient completing two courses of therapy without experiencing a grade 4 or 5 non-hematologic toxicity.

SECONDARY OUTCOMES:
Toxicity profile of patients with SMN treated with one or two courses of CPX-351 | 30 days after completion of one or two courses of chemotherapy
  We will define categories for toxicity events and for each category we will determine the highest grade experienced by each patient. We will then report the number of patients with each grade in each category.
Biologic correlates of response in patients with SMN after one or two courses of CPX-351 | Day 22 for the first cycle and day 36-42 after the second cycle
  We will use logistic regression modeling explore biologic correlates as predictors of response. For genomic associations, we will use false discovery rate methods to address multiple testing.
Overall (OS) survival of patients who received one or two courses of CPX-351 followed by HSCT | 3 years from study entry
  We will use the Kaplan-Meier method to estimate overall survival. We define OS as the time elapsed from protocol enrollment to death and censor times of living patients at last follow-up.
Event-free survival (EFS) of patients who received one or two courses of CPX-351 followed by HSCT | 3 years from study entry
  We will use the Kaplan-Meier method to estimate event-free survival. We define EFS as the time elapsed from protocol enrollment to death, relapse, discontinuation of therapy due to excessive toxicity or resistant disease, or development of an additional malignancy and censor times for patients free of these events at last follow-up.
The impact of transplant on patients who received one or two courses of CPX-351 followed by HSCT | 3 years from study entry
  To explore the impact of transplant, we will fit Cox models with transplant as a time-dependent covariate.

CONTACTS AND LOCATIONS:
Overall Officials: Raul C. Ribeiro, MD, Principal Investigator — St. Jude Children's Research Hospital; Marcin Wlodarski, MD, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT05656248/Prot_SAP_000.pdf
  • Informed Consent Form (2025-06-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT05656248/ICF_001.pdf